CLINICAL TRIAL: NCT00185731
Title: A Phase II Study of Atorvastatin in Patients With Low Grade or Refractory Non-Hodgkin's Lymphoma
Brief Title: Phase 2 Study of Atorvastatin Safety and Antitumor Effects in Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dean Felsher (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); Damon Runyon Cancer Research Foundation (Other); Burroughs Wellcome (Industry)
Responsible Party: Sponsor-Investigator, Dean Felsher, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13683; 4328-07 (Other: Damon Runyon Cancer Research Foundation); 95140 (Other: Stanford University Alternate IRB Approval Number); LYMNHL0020 (Other: OnCore)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Leukemia; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 80 mg Atorvastatin (Experimental): Atorvastatin, 80 mg tablet, will be taken orally by the patient daily, beginning on study day 1.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 80 mg orally once daily
  Other Names: Lipitor

SUMMARY:
This is an approach which can inflict significant toxicity. An alternative is to block expression of oncogenes which are over-expressed only in cancer cells, a therapeutic approach which could reduce toxicity to the host while maximizing destruction of the oncogene-dependent malignant cells.

DETAILED DESCRIPTION:
Atorvastatin has been shown to decrease levels of active oncogenes in preclinical studies with murine and human lymphoma cell lines, and administration of statins leads to shrinkage of lymphoma in murine models. Therefore, it may be possible for atorvastatin to decrease levels of active oncogenes in human lymphomas. Further, upon decrease in levels of active oncogenes, human lymphomas may regress. Atorvastatin is a commonly prescribed drug for hypercholesterolemia: targeting the 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase enzyme may also be a way to decrease activation of oncogenes in human lymphoma, with minimal toxicity. For human low grade non-Hodgkin lymphoma, no curative treatment is available; therefore new, non-toxic and targeted therapies are sought for this disease.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Disease criteria: Confirmed by Stanford Pathology to be one of the following Non-Hodgkin's Lymphoma (NHL) subtypes:

  * Chronic lymphocytic leukemia /small lymphocytic lymphoma (CLL/SLL)
  * Extranodal marginal zone B-cell lymphoma
  * Nodal marginal zone B-cell lymphoma
  * Splenic marginal zone B-cell lymphoma
* Treatment criteria

  * Untreated: watchful waiting currently appropriate (includes CLL stage 0) o OR
  * Prior treatment: watchful waiting currently appropriate o OR
  * Refractory disease
* Staging within 4 weeks prior to enrollment (SLL, marginal zone lymphoma)

  * CT chest (date)
  * CT abdomen (date)
  * CT pelvis (date) OR
* Staging within 4 weeks prior to enrollment (CLL: CT not required)

  * Total white blood cell count (WBC) (Value) (date)
  * Absolute lymphoma cell count (ALC) (Value) (date)
  * Measurable disease (Site) (Size) OR
  * CLL (only): elevated absolute lymphoma cell count
* Disease amenable to biopsy (must check at least one):

  * Circulating tumor cells
  * Positive bone marrow
  * Palpable involved site (such as lymph node) measuring > 1.5 cm
* Eastern Cooperative Oncology Group performance status <2 (Karnofsky >60)
* Life expectancy of greater than 3 months
* Patients must have adequate organ and marrow function

  * Absolute neutrophil count > 1,000/uL
  * Platelets > 30,000/uL
  * Total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ratio < 2.5 x institutional upper limit of normal
  * Creatinine within normal institutional limits OR creatinine clearance > 60 mL/min/1.73 m² for patients with creatinine levels above institutional normal.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Women of child-bearing potential must have negative BetaHCG at enrollment

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Not recovered from adverse events due to agents administered more than four weeks earlier
* Has stable low grade lymphoma has had rituximab within 3 months Patient with relapsed or refractory disease has had rituximab within 1 month
* Not recovered from adverse events due to surgery performed 4 weeks earlier
* Receiving any other investigational agent. Known brain metastases
* Taken any statin within the past 6 months prior to enrollment in the trial
* Currently abuses alcohol
* Currently takes cyclosporin or gemfibrozil Patient has a prior history of rhabdomyolysis
* Has uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant: Patients are not excluded if they are breastfeeding at the time of enrollment, but breastfeeding should be discontinued if the mother is treated with atorvastatin.
* HIV-positive patients receiving combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Felsher, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin: Atorvastatin, 80mg tablet, orally once daily.
Period: Overall Study
Arm/Group | Atorvastatin
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Not Eligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Atorvastatin
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 3
Histology [Count of Participants; unit: Participants]
  Small Lymphocytic Lymphoma | 16
  Follicular Lymphoma | 6
  Marginal Zone B-Cell Lymphoma | 2
  Splenic Marginal Zone B-Cell Lymphoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Apoptosis
Description: Expressed as the number of participants whose tumor cells showed an increase in apoptosis during atorvastatin treatment
Time Frame: 1 year
Population: 24 participants had tumors sampled for primary endpoint as per protocol. However, 1 withdrew, and only 22 of remaining participants had adequate tumor samples for analysis of apoptosis at baseline and at subsequent time points.
Measure: Count of Participants; unit: Participants
Groups:
- Atorvastatin: Atorvastatin, 80mg tablet, was taken orally by the patient daily, beginning on study day 1.
  Atorvastatin: 80 mg orally once daily
Arm/Group | Atorvastatin
Number analyzed (Participants) | 22
Participants | 7

2. Secondary Outcome: Correlation of Tumor Apoptosis to Clinical Response
Description: The validity of tumor apoptosis as a biologic endpoint was assessed by correlation to clinical response. A correlation substantially less than 1 is interpreted as a poor correlation, while a correlation near +1 or -1 is interpreted as a strong correlation.
Time Frame: 1 year
Population: 24 participants had tumors sampled for primary endpoint as per protocol. However, 1 withdrew and 1 had an inadequate tumor samples for analysis, leaving only 22 remaining participants for analysis of apoptosis at baseline and at subsequent time points.
Measure: Number; unit: Pearson Correlation Coefficient
Groups:
- 80 mg: Atorvastatin, 80 mg tablet, was taken orally by the patient daily, beginning on study day 1.
  Atorvastatin: 80 mg orally once daily
Arm/Group | 80 mg
Number analyzed (Participants) | 22
Pearson Correlation Coefficient | -0.26

3. Secondary Outcome: Atorvastatin Toxicity
Description: Assessed as the number of study participants with atorvastatin-related serious adverse events (SAEs).
Time Frame: 1 year
Population: All study participants who received atorvastatin
Measure: Count of Participants; unit: Participants
Groups:
- 80 mg Atorvastatin: Atorvastatin, 80 mg tablet, was taken orally by the patient daily, beginning on study day 1.
  Atorvastatin: 80 mg orally once daily
Arm/Group | 80 mg Atorvastatin
Number analyzed (Participants) | 24
Participants | 4

ADVERSE EVENTS:
Description: 1 participant found not to be eligible and was not analyzed
Arm/Group | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 4/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=24)
Diarrhoea (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Mood alteration - Anxiety (Psychiatric disorders) | 1
Pain - Abdominal NOS (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=24)
elevated SGOT (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 5
elevated SGPT (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 6
elevated alk phos (alkaline phosphatase) (Hepatobiliary disorders) | 3
infection (Infections and infestations) | 4 — (upper respiratory)
nausea (Gastrointestinal disorders) | 3
hematoma (Musculoskeletal and connective tissue disorders) | 2
low platelets (Blood and lymphatic system disorders) | 1
elevated platelets (Blood and lymphatic system disorders) | 1
constipation (Gastrointestinal disorders) | 2
diaphoresis (General disorders) | 1 — night sweats (1)
pain (General disorders) | 13 — myalgia (2), pain NOS (2), leg cramps (2), back pain (1), leg pain (1), right upper quadrant pain (1), toe pain (1), abdominal pain (1), headache (1), neurologic pain (1)
diarrhea (Gastrointestinal disorders) | 4
fatigue (General disorders) | 1
hyperbilirubinemia (Hepatobiliary disorders) | 2
anorexia (Gastrointestinal disorders) | 1
bloating (Gastrointestinal disorders) | 1
palpitation (Cardiac disorders) | 1
vomiting (Gastrointestinal disorders) | 1
vasculitis (Vascular disorders) | 1
bruising (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No